CLINICAL TRIAL: NCT01677689
Title: A Prospective, Randomized, Double-blind, Parallel, Placebo-controlled, Multi-center Study to Investigate the Efficacy and Safety of Apomivir® in Relieving Influenza Symptoms
Brief Title: Study to Investigate the Efficacy and Safety of Apomivir®
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Far East Bio-Tec Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QCR09032
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Influenza
Keywords: oral temperature; respiratory symptom; cough; nasal obstruction; sore throat; fever
MeSH Terms: conditions — Influenza, Human; Signs and Symptoms, Respiratory; Cough; Nasal Obstruction; Pharyngitis; Fever

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Placebo Comparator): Placebo 1 capsule twice daily. All subjects will be treated for 5 days, and all drugs should be taken orally after meal
  Interventions: Drug: Placebo
- Study Group (Experimental): Apomivir® 1 capsule twice daily. All subjects will be treated for 5 days, and all drugs should be taken orally after meal.
  Interventions: Drug: Apomivir®

INTERVENTIONS:
Drug: Apomivir® — Study Group: Apomivir® 1 capsule twice daily. All subjects will be treated for 5 days, and all drugs should be taken orally after meal.
  Other Names: FE-L-APO(drug substance)
  Arms: Study Group
Drug: Placebo — Control Group: Placebo 1 capsule twice daily. All subjects will be treated for 5 days, and all drugs should be taken orally after meal.
  Arms: Control Group

SUMMARY:
Apomivir® is extracted from a proprietary spirulina strain, FEM-101, a kind of blue cyanobacterium with patented freeze-thaw lysis and extraction method. According to the preclinical studies, Apomivir® have been proven to have excellent broad-spectrum anti-viral ability, especially for seasonal influenza viruses (Influenza virus A and B) that may cause illness, paralysis and even death, especially in children and elderly people. This phase II study is designed to evaluate the efficacy and safety of Apomivir® (120 mg b.i.d.) in subjects with seasonal influenza.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, parallel, placebo-controlled, multi-center study. Approximately 196 subjects with fever defined as body temperature >= 38˚C, with at least one respiratory symptom and one other constitutional symptom will be invited into this study to target 156 evaluable subjects. A nasopharyngeal/throat swabs rapid test for influenza A and B will be conducted and only subjects with positive results could be recruited. All eligible subjects will be randomized to one of the following treatment group in a 1:1 ratio.

Study Group: Apomivir® 1 capsule (120 mg/cap) twice daily for 5 days Control Group: Placebo 1 capsule twice daily for 5 days A pack of acetaminophen (500 mg) will be provided at enrollment. All flu symptom relief agents could be used only for rescue use of persistent fever or flu symptoms (>= 24 hours). A digital thermometer and diary card will be dispensed at baseline (Day 1). Subjects will be instructed to complete the body temperature record, and daily record regarding the severity of their influenza symptoms and the level of interference on daily activity. The monitoring frequency will be twice daily (after drug administration) from Day 1 to Day 5, and cut down to once daily until Day 29 or completed cure (defined as remission of all flu symptoms and interferences). Treatment failure is defined as secondary illnesses, antibiotic use and hospitalization due to disease progression.

For safety and efficacy assessments, all subjects should return on Day 3, 6 and 15. For subjects who are not completely cured before Day 15 (Visit 4), further therapy will be conducted and they should return on Day 29; for those who are completely cured, only a telephone follow-up will be conducted on Day 29.

The severity of fever will be scored using a 4-point scale:

0 = < 37.2°C

1. = >= 37.2 to < 38.0°C
2. = >= 38.0 to < 39.0°C
3. = >= 39.0 °C

Other influenza symptoms (such as cough, nasal obstruction, sore throat, fatigue, headache and myalgias) will also be assessed using a 4-point scale:

0 = none,

1. = mild,
2. = moderate,
3. = severe

The level of interference on daily activities (including running, lifting heavy objects, participating in strenuous sports, moderate activities), such as moving a table, pushing a vacuum cleaner, bowling, or playing golf, lifting or carrying groceries, climbing several flights of stairs, climbing one flight of stairs, bending, kneeling, or stooping, walking more than a mile, walking several blocks, walking one blocks, and bathing or dressing yourself, will be assessed according to a 3-point scale

0 = no, no limited

1. = yes, limited a little
2. = yes, limited a lot

Confirmatory tests for infective virus strain, real-time RT-PCR and viral culture will be conducted at baseline. In the following study visits, real-time RT-PCR will be performed to measure the influenza viral load/titer in nasopharyngeal/throat swabs specimen. For those who have been completely cured prior to Day 15, the real-time RT-PCR assessment could be omitted on Day 29. All subjects enrolled will be followed until the end of study, but only subjects with influenza PCR or viral culture positive could be evaluable population.

ELIGIBILITY:
1. Main inclusion criteria:

1. Females and males aged between 20 and 65
2. Presumptive diagnosis of influenza based on the following clinical characteristics:

   * Present at least one respiratory symptom (e.g. cough, nasal obstruction, sore throat) and at least one constitutional symptom other than fever (e.g. fatigue, headache, myalgias) of less than 48-hour duration
   * Positive for influenza A or B (nasopharyngeal/throat swab - rapid test)
3. Able and willing to comply with the study procedure and give written informed consent

2. Main exclusion criteria:

1. Female who is pregnant/lactating or planning to be pregnant, or female of childbearing potential* who is not using medically recognized method of contraception

   * Other than those who have been surgically sterilized (defined as having undergone hysterectomy or bilateral oophorectomy or bilateral salpingectomy; tubal ligation alone is not considered sufficient) or one year post-menopausal
2. Subject with chronic pulmonary diseases or critical condition or already developed severe respiratory distress with hypoxaemia on presentation
3. Subject with a history of non-febrile convulsions, neuromuscular disorders or cognitive dysfunction that may compromise respiratory secretions, or who are currently receiving anticonvulsive agents
4. Subject with clinically important illness, malignancies, systemic infection, other medical or psychiatric condition which places the subject at unacceptable risk to participate in the study or confounds the ability to interpret data from the study
5. Subject with significant abnormal laboratory findings (hemoglobin level < 9.0 g/dL, WBC < 4000/mm3, platelet count < 100,000/mm3, ALT or AST > 2.5 x upper limit of normal (ULN), or estimated creatinine clearance < 30 mL/min within 4 weeks prior to baseline)
6. Subject who are currently receiving immunosuppressive therapy,
7. Subject has taken daily supplement(s) containing blue agar within 1 month prior to screening, or any other medication that may affect the study results
8. Known hypersensitivity to any ingredients in Apomivir® or other blue agar
9. Use of any investigational product within 1 month prior to screening

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2026-05-31 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety profile of Apomivir® treatment (120 mg b.i.d.). | from day1 to day 29, the entire treatment period and follow-up period.
  Safety endpoints:
  1. Change in laboratory data
  2. Adverse events
  3. Serious adverse events (SAE)
To evaluate the time to resolution of influenza symptoms defined as all flu symptom scores ≤ 1 after initiation of study treatment. | from day 1 to day 29, depends on the time to sympton resolution of individual subjects.
  The time to resolution of influenza symptom is defined as the duration from the study drug initiation to all flu symptom scores ≤ 1. Subject who is withdrawn prior to the resolution of influenza symptom is censored at the last known time point.

SECONDARY OUTCOMES:
Change in virus titer. | Day 3, 6 compared to baseline (Day 1)
  To evaluate the change in virus titer assessed by real-time RT-PCR15.
Time to achieve afebrile | after initiation of study treatment
  Time to bring down a fever (oral temperature < 37.2˚C)
Severity of influenza symptom score during study period | twice daily from Day 1 to Day 6 and once daily until Day 29 or completely cured
  All subjects should complete the diary card twice daily from Day 1 to Day 6 and cut down to once daily until Day 29 or completely cured.
Level of interference on daily activity and time to alleviation of the interference during study period | twice daily from Day 1 to Day 6 and once daily until Day 29 or completely cured
  All subjects should complete the diary card twice daily from Day 1 to Day 6 and cut down to once daily until Day 29 or completely cured.
Proportion of rescue medication used for fever or influenza symptoms during study period | twice daily from Day 1 to Day 6 and once daily until Day 29 or completely cured
  All subjects should complete the diary card twice daily from Day 1 to Day 6 and cut down to once daily until Day 29 or completely cured.
Proportion and time to treatment failure during study period | from day 1 to day 29, including treatment period and follow-up period
  Proportion and time to treatment failure (including secondary illnesses, antibiotic use and hospitalization due to disease progression) during study period

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Wen Hang, MD, Principal Investigator — China Medical University Hospital; YI-HSIANG CHEN, Study Director — Far East Bio-Tec Co., Ltd
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

REFERENCES:
- [Background] Lynch G, Low L, Li S, Sloane A, Adams S, Parish C, Kemp B, Cunningham AL. Sulfated polyanions prevent HIV infection of lymphocytes by disruption of the CD4-gp120 interaction, but do not inhibit monocyte infection. J Leukoc Biol. 1994 Sep;56(3):266-72. doi: 10.1002/jlb.56.3.266. PMID 7521897
- [Background] Shih CM, Cheng SN, Wong CS, Kuo YL, Chou TC. Antiinflammatory and antihyperalgesic activity of C-phycocyanin. Anesth Analg. 2009 Apr;108(4):1303-10. doi: 10.1213/ane.0b013e318193e919. PMID 19299804
- [Background] Gonzalez R, Rodriguez S, Romay C, Ancheta O, Gonzalez A, Armesto J, Remirez D, Merino N. Anti-inflammatory activity of phycocyanin extract in acetic acid-induced colitis in rats. Pharmacol Res. 1999 Jan;39(1):55-9. PMID 10366332
- [Background] Shih SR, Tsai KN, Li YS, Chueh CC, Chan EC. Inhibition of enterovirus 71-induced apoptosis by allophycocyanin isolated from a blue-green alga Spirulina platensis. J Med Virol. 2003 May;70(1):119-25. doi: 10.1002/jmv.10363. PMID 12629652
- [Background] Reagan-Shaw S, Nihal M, Ahmad N. Dose translation from animal to human studies revisited. FASEB J. 2008 Mar;22(3):659-61. doi: 10.1096/fj.07-9574LSF. Epub 2007 Oct 17. PMID 17942826
- See also: The drug substance of the IP is the same with a marked nutrition supplement. And this is the official product page of the marked nutrition supplement. — http://www.febico.com.tw